CLINICAL TRIAL: NCT06789848
Title: Phase II Basket Trial of Ligufalimab (AK117) and Cadonilimab (AK104) in Advanced Hepatobiliary Cancers
Brief Title: Ligufalimab and Cadonilimab in Advanced Liver Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Akesobio (Industry); Josephine Hughes Sterling Foundation (Unknown)
Responsible Party: Principal Investigator, David Hsieh, Assistant Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-15224; STU-2024-1210
Record Dates: First submitted 2025-01-21; First posted 2025-01-23 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Advanced Hepatocellular Carcinoma; Refractory Hepatocellular Carcinoma; Biliary Tract Cancer
Keywords: liver; other digestive organs
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: Hepatocellular carcinoma (HCC) / Liver Cancer (Experimental): Ligufalimab and Cadonilimab are given via intravenous (through the veins) infusion in the clinic. Each clinic visit will last 4-5 hours. Infusions of study drugs will be given on the first day of every 21-day cycle. Study medications will continue if evaluations show that disease has not gotten worse.
  Interventions: Drug: Ligufalimab; Drug: Cadonilimab
- Cohort B: Bile duct cancer (Experimental): Ligufalimab and Cadonilimab are given via intravenous (through the veins) infusion in the clinic. Each clinic visit will last 4-5 hours. Infusions of study drugs will be given on the first day of every 21-day cycle. Study medications will continue if evaluations show that disease has not gotten worse.
  Interventions: Drug: Ligufalimab; Drug: Cadonilimab

INTERVENTIONS:
Drug: Ligufalimab — Ligufalimab (AK117) 45 mg/kg IV over 120 minutes on Day 1 every 3 weeks
Drug: Cadonilimab — Cadonilimab (AK104) 10 mg/kg IV over 60 minuets at least 30 minutes after Ligufalimab on Day 1 every 3 weeks

SUMMARY:
The goal of this clinical trial is to find out if the combination of Ligufalimab and Cadonilimab are effective in treating advanced hepatobiliary cancers that have failed prior therapy.

DETAILED DESCRIPTION:
The study is an open-label, non-randomized, phase II basket therapeutic clinical trial. To determine the objective response rate of combination ligufalimab and cadonilimab in refractory and advanced hepatocellular carcinoma and biliary tract cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of specific disease -Cohort A (HCC): Patient must have a diagnosis confirmed by histology or clinically by the American Association for the Study of Liver Diseases (AASLD) criteria in patients with cirrhosis. Known fibrolamellar HCC will be excluded.

   * Cohort B (BTC, biliary tract cancers): Patients must have histologically confirmed biliary tract cancer (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gall bladder cancers). Patients with combined HCC-cholangiocarcinoma may be enrolled in Cohort B.
2. Locally advanced or metastatic disease

   * Patients with locally advanced or metastatic disease must have disease deemed not amenable to surgical and/or locoregional therapies or patients who have progressed following surgical and/or locoregional therapies.
   * Measurable disease, as defined as lesions that can accurately be measured in at least one dimension according to RECIST version 1.1 at least 1 cm with contrast enhanced dynamic imaging (magnetic resonance imaging or computed tomography).
3. Refractory to or relapsed after prior anti-PD-1/L1 antibody therapy. May have received anti-PD-1/L1 monotherapy or combination therapy as any line of therapy including in the neoadjuvant or adjuvant setting. Patients who discontinued prior immune checkpoint inhibitor treatment due to a high-grade toxicity (Grade 4) are not eligible.
4. For patients in cohort A who do not have a clinical diagnosis of HCC according to the AASLD criteria, formalin-fixed, paraffin-embedded (FFPE) tumor diagnostic tissue samples must have been obtained within 4 years from the time of consent. Baseline tissue will be requested any time after consent. It is strongly recommended that tissue is obtained from standard-of-care biopsies confirming progression of disease on prior therapy so that the patient has not received any intervening systemic anti-cancer treatment from the time that the baseline tissue was obtained.
5. Prior locoregional therapy is allowed provided the following are met: 1) at least 2 weeks since prior locoregional therapy including surgical resection, chemoembolization, radiotherapy, or ablation; 2) target lesion has increased in size ≥25% since the cessation of locoregional therapy or the target lesion was not treated with locoregional therapy. Patients treated with palliative radiotherapy for symptoms will be eligible as long as the target lesion is not the treated lesion and radiotherapy will be completed at least 2 weeks prior to study drug administration.
6. Age ≥ 18 years
7. Child-Pugh Score A or B7 (only applicable for Cohort A)
8. ECOG Performance score of 0-1
9. Adequate organ and marrow function (without chronic, ongoing growth factor support or transfusion in the last 2 weeks) as defined below:

   -Platelet count ≥ 50,000/mm3

   -Hgb ≥ 9 g/dl

   -Absolute neutrophil ≥ 1,000 cells/mm3

   -Total bilirubin ≤ 3 mg/ml (This will not apply to subjects with Gilbert's syndrome who have persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis, or patients with hyperbilirubinemia secondary to distal malignant obstruction where endoscopic, surgical, or percutaneous bypass/stenting has been attempted. Such patients may be enrolled based in consultation with the principal investigator)

   -INR ≤ 2

   -AST, ALT ≤ 5 times ULN
   * Calculated creatinine clearance (CrCl) ≥ 40 mL/min. CrCl can be calculated using the Cockroft-Gault method.
   * Albumin ≥ 2.0 g/dl
10. All men, as well as women of child-bearing potential, defined as not surgically sterilized and between menarche and 1-year post menopause, must agree to use highly effective contraception methods (hormonal or barrier method of birth control or abstinence) 4 weeks prior to study entry, for the duration of study participation, and for 120 days after the last dose of ligufalimab or cadonilimab.

Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  11. Women of child-bearing potential must have a negative serum pregnancy test at screening.

  12. Subjects are eligible to enroll if they have non-viral-HCC, or if they have HBV-HCC, or HCV-HCC defined as follows:

  1) HBV-HCC: Hepatitis B subjects will be allowed if they meet the following criteria: On antiviral therapy for HBV. Subjects who are anti-HBc (+), negative for HBsAg, negative for anti-HBs, and have an HBV viral load under 100 IU/mL do not require HBV anti-viral prophylaxis.

  2) HCV-HCC: Active or resolved HCV infection as evidenced by detectable HCV RNA or antibody. Patients who have failed HCV therapy as evidenced by detectable HCV RNA will be eligible. Subjects with chronic infection by HCV who are treated (successfully or treatment failure) or untreated are allowed on study.

  13. Ability to understand and the willingness to sign a written informed consent.

  14. Willing and able to comply with the requirements and restrictions in this protocol.

  15. Patients who have received the vector, protein subunit, or nucleic acid COVID-19 vaccines are eligible to enroll.

Exclusion Criteria:

1. Prior liver transplant.
2. Known human immunodeficiency virus (HIV) positive (testing not required).
3. Use of any live vaccines against infectious diseases within 28 days of first dose of study drug administration.
4. History of trauma or major surgery within 28 days prior to the first dose of study drug administration. (Tumor biopsy or placement of central venous access catheter (eg, port or similar) is not considered a major surgical procedure).
5. Underlying medical conditions that, in the investigator's opinion, will make the administration of study drugs hazardous, including but not limited to:

   * Interstitial lung disease, including history of interstitial lung disease or non infectious pneumonitis (lymphangitic spread of cancer is not disqualifying),
   * Active viral, bacterial, or fungal infections requiring parenteral treatment within 14 days of the initiation of study drugs,
   * Clinically significant cardiovascular disease,
   * A condition that may obscure the interpretation of toxicity determination or AEs,
   * History of prior solid-organ transplantation.
6. Hypersensitivity to IV contrast; not suitable for pre-medication.
7. Any active autoimmune disease or a documented history of autoimmune disease or syndrome that required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs), except for vitiligo or resolved childhood asthma/atopy.

   * Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
   * Participants with asthma who require intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections will not be excluded from this study. Participants on chronic systemic corticosteroids will be excluded from the study.
8. Known history of active bacillus tuberculosis.
9. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone equivalent) or other immunosuppressive medications within 14 days of study administration. Inhaled or topical steroids and adrenal replacement doses ≤10 mg/day prednisone equivalents are permitted in the absence of autoimmune disease.
10. Patients who discontinued prior immune checkpoint inhibitor treatment due to Grade ≥ 3 or Grade 2 serious toxicity (i.e., pneumonitis, uveitis, neurological symptoms, cardiac toxicity, etc.) immune-related adverse events.
11. Known severe hypersensitivity reactions to monoclonal antibodies (≥Grade 3).
12. Prior malignancy that required systemic treatment within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or prostate cancer.
13. Prisoners or subjects who are involuntarily incarcerated.
14. If a participant has symptomatic or clinically active brain metastases including leptomeningeal disease, they must be excluded if:

    * Has evidence of progression by neurologic symptoms
    * Has metastatic brain lesions that require immediate intervention.
    * Has carcinomatous meningitis, regardless of clinical stability
15. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after contraception and until the termination of gestation, confirmed by a positive hCG laboratory test.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Has significant dementia or other mental condition that precludes the participant's ability to consent to the study.
18. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of study drugs.
19. Known hypersensitivity to recombinant proteins, or any excipient contained in the study drug formulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response rate of combination ligufalimab and cadonilimab | Study treatment will continue until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  To determine the best objective response rate assessed by RECIST guidelines (version 1.1) of combination ligufalimab and cadonilimab in patients with advanced hepatobiliary cancers previously exposed to anti-PD-1/L1 antibody treatments.

SECONDARY OUTCOMES:
Overall survival of combination ligufalimab and cadonilimab | Study treatment will continue until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  To determine the overall survival rate of response of combination ligufalimab and cadonilimab compared to historical controls assessed by RECIST guidelines (version 1.1)
Progression-free survival of combination ligufalimab and cadonilimab | udy treatment will continue until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  To determine the progression-free survival rate of response of combination ligufalimab and cadonilimab compared to historical controls assessed by RECIST guidelines (version 1.1)
Duration of response of combination ligufalimab and cadonilimab | Study treatment will continue until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  To determine the duration of response of combination ligufalimab and cadonilimab compared to historical controls assessed by RECIST guidelines (version 1.1)
Overall safety profile of combination ligufalimab and cadonilimab. | Study treatment will continue until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  Safety profile of combination ligufalimab and cadonilimab will be measured by the number of participants with Adverse Events (AEs) (serious / non-serious) as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: David Hsieh, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No